CLINICAL TRIAL: NCT00137202
Title: A Pilot Study to Determine the Pruritic Benefits of Ondansetron Versus Diphenhydramine in Burn Patients Undergoing Wound Healing
Brief Title: Post Burn Pruritus Study in Patients Undergoing Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: USAISR
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-04-006
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Itching
Keywords: pruritus; burn wound
MeSH Terms: conditions — Pruritus; Burns | interventions — Ondansetron; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Active Comparator)
  Interventions: Drug: Ondansetron (Zofran); Drug: Diphenhydramine (Benadryl)

INTERVENTIONS:
Drug: Ondansetron (Zofran)
Drug: Diphenhydramine (Benadryl)

SUMMARY:
The purpose of this study is to see if a drug called ondansetron (Zofran) controls itching from healing burn wounds as well or better than the usual drug used, diphenhydramine (Benadryl).

DETAILED DESCRIPTION:
A clear mechanism or cause for pruritus in patients recovering from burn has not been delineated.

While the exact mechanisms/pathways for itching are currently unclear, histamine antagonism appears to be the most popular treatment. Whether histamine antagonism works predominantly via peripheral inhibition or central sedation is uncertain. By treating another intermediary in the pruritus cascade, it may be possible that an alternate treatment could be used while eliminating some of the unwanted side effects of antihistamine at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Males or females; 18 years or older.
* Seen in the United States Army Institute of Surgical Research (USAISR) Burn Clinic with healing burn wounds of any percent (%) of total body surface area (TBSA) causing pruritus
* Stable medical condition
* Negative pregnancy test and not nursing
* Able to indicate status of pruritus on a numeric scale
* Able to understand and read English

Exclusion Criteria:

* Unstable medical condition as determined by attending burn surgeon
* Prisoner
* History of allergic reaction to serotonin inhibitors or diphenhydramine
* Pregnant or lactating
* Unable to verbalize pruritus intensity scale
* Unable to understand or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Ondansetron will have a greater ability to control pruritus in burn patients who are undergoing wound healing when compared to the standard of care, diphenhydramine. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Gross, MD, Principal Investigator — Wilford Hall Medical Center, Lackland AFB, San Antonio, TX; Steven E Wolf, MD, Study Director — US Army Institute of Surgical Research, Fort Sam Houston, TX
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Matheson JD, Clayton J, Muller MJ. The reduction of itch during burn wound healing. J Burn Care Rehabil. 2001 Jan-Feb;22(1):76-81; discussion 75. doi: 10.1097/00004630-200101000-00017. PMID 11227690